CLINICAL TRIAL: NCT01177163
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-28431754 in Type-2 Diabetes Mellitus Subjects Not Optimally Controlled (A1C >=7.0%) on Fixed Doses of Insulin Therapy
Brief Title: A Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Study of JNJ-28431754 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR014881
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes mellitus; Canagliflozin; JNJ-28431754; Insulin; Pharmacokinetic; Pharmacodynamic; SGLT-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 001 (Other): Placebo one placebo capsule once daily for 3 days immediately prior to randomization to double-blind treatment with JNJ 28431754 or placebo
  Interventions: Drug: Placebo
- 002 (Experimental): JNJ 28431754 100 mg/placebo one 100-mg capsule of JNJ-28431754 or placebo once-daily for 4 weeks
  Interventions: Drug: JNJ 28431754 100 mg/placebo
- 003 (Experimental): JNJ 28431754 300 mg/placebo one 300-mg capsule of JNJ-28431754 or placebo twice-daily for 4 weeks
  Interventions: Drug: JNJ 28431754 300 mg/placebo

INTERVENTIONS:
Drug: Placebo — one placebo capsule once daily for 3 days immediately prior to randomization to double-blind treatment with JNJ 28431754 or placebo
  Arms: 001
Drug: JNJ 28431754 300 mg/placebo — one 300-mg capsule of JNJ-28431754 or placebo twice-daily for 4 weeks
  Arms: 003
Drug: JNJ 28431754 100 mg/placebo — one 100-mg capsule of JNJ-28431754 or placebo once-daily for 4 weeks
  Arms: 002

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacodynamic effects and pharmacokinetic characteristics of JNJ-28431754 after multiple dosing in patients with Type 2 Diabetes Mellitus who are on a stable dose of insulin.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), double-blind (neither the patient or the study doctor will know the name of the assigned treatment), parallel-group (each group of patients will be treated at the same time) to determine the safety, tolerability, pharmacokinetics (PK) (how drugs are absorbed in the body, how they are distributed within the body and how they are removed from the body over time) and the pharmacodynamics (PD) (the action or effects a drug has on the body) of oral (taken by mouth) doses of JNJ 28431754 taken once or twice daily compared to placebo (treatment identical in appearance to JNJ-2843174 but contains no active drug) in patients with Type 2 Diabetes Mellitus (T2DM) who are receiving therapy with a fixed-dose regimen of insulin. Two groups of 14 patients will be studied; one group will receive JNJ-2843174 (100 mg) or placebo once daily for 4 weeks and the other group will receive JNJ-2843174 (300 mg) or placebo twice daily for 4 weeks. In the 3 days immediately prior to the beginning of the 4-week treatment period, all patients will take a single oral dose of placebo once daily and have blood and urine samples collected for laboratory testing. During the study, all patients will be allowed to continue on their normal medication regimen of insulin and other allowed anti-diabetic medications. On selected days during the study, patients will be required to stay overnight at the study center to have study drug administered and/or to have blood and urine samples collected for laboratory testing. During the study, if patients experience worsened glycemia (blood sugar), rescue therapy with additional insulin of the same type but at a higher dose may be initiated by the Investigator if medically appropriate. During the study, patients will be monitored for safety by review of adverse events and results from laboratory tests, 12-lead electrocardiograms (ECGs), vital signs measurements, body weight, physical examinations, and self-monitored blood glucose (SMGB) measurements. Unless otherwise specified, study drug will be taken orally (by mouth) after an overnight fast for at least 8 hours followed by a meal within 10 minutes; for twice daily dosing, the evening dose will be taken just prior to the evening meal (dinner). All patients will take one placebo capsule once daily for 3 days immediately prior to randomization. After randomization, patients will take JNJ-28431754 (100 mg) or placebo once daily or JNJ-28431754 (300 mg) or placebo twice daily for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with T2DM for at least 6 months prior to study screening
* Be on stable insulin regimens at the time of screening
* Have a stable weight (ie, no change more than 5% in the 3 months prior to screening)
* Have a glycosylated hemoglobin (A1C) of >=7% and <=10.5% at study screening

Exclusion Criteria:

* Have history of Type 1 diabetes mellitus, secondary forms of diabetes, diabetic ketoacidosis, pancreas or beta cell transplantation
* Have a known history of more than 2 severe hypoglycemic episodes as defined by the protocol within the past year
* Have history of, or currently active, significant illness as determined by the Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-05; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who need to decrease insulin dosage from prestudy dosage levels because of hypoglycemia | From time of signed informed consent (Days -52 to -32) through to the end of the study (Days 34 to 39) or at the time of early withdrawal
The number of patients with specific treatment-emergent adverse events | From time of signed informed consent (Days -52 to -32) through to the end of the study (Days 34 to 39) or at the time of early withdrawal
The number of patients with symptomatic hypoglycemia and severe hypoglycemia | From time of signed informed consent (Days -52 to -32) through to the end of the study (Days 34 to 39) or at the time of early withdrawal

SECONDARY OUTCOMES:
Plasma concentrations and pharmacokinetics parameters for JNJ 28431754 | At protocol-specified timepoints from Day 1 (pre-dose) to Day 29
Plasma glucose concentration-time profiles (pharmacodynamics parameter) | At protocol specified timepoints on Day -1, Day 1, and Day 27
Change in urine glucose excretion (pharmacodynamics parameter) | At protocol specified timepoints on Day -1, Day 1, and Day 27

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (2):
- United States (2):
  - Chula Vista, California
  - San Antonio, Texas

REFERENCES:
- See also: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-28431754 in T2DM Subjects not Optimally Controlled (HbA1c: ≥7.0%) on Fixed Doses of Insulin Therapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=787&filename=CR014881_CSR.pdf